CLINICAL TRIAL: NCT05852782
Title: Effects of Narrowband and Broadband Light on Choroidal Thickness and Melanopsin-driven Pupil Response
Brief Title: Effects of Light on the Choroid and Pupil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001524
Record Dates: First submitted 2023-04-27; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2019-01

CONDITIONS: Emmetropia; Myopia
MeSH Terms: conditions — Myopia | interventions — Phototherapy; Darkness

STUDY DESIGN:
Intervention Model Description: All subjects will participate in four conditions on separate days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Light exposure broadband (Experimental): Participants will be exposed to indoor levels of light that appear colorless for one hour
  Interventions: Other: White Light therapy
- Light exposure long wavelength (Experimental): Participants will be exposed to indoor levels of light that appear red for one hour
  Interventions: Other: Red light therapy
- Light exposure short wavelength (Experimental): Participants will be exposed to indoor levels of light that appear blue for one hour
  Interventions: Other: Blue light therapy
- Light exposure darkness (Experimental): Participants will be exposed to darkness for one hour
  Interventions: Other: Darkness

INTERVENTIONS:
Other: White Light therapy — Participants will be exposed to broadband light for one hour
  Arms: Light exposure broadband
Other: Blue light therapy — Participants will be exposed to blue light for one hour
  Arms: Light exposure short wavelength
Other: Red light therapy — Participants will be exposed to re light for one hour
  Arms: Light exposure long wavelength
Other: Darkness — Participants will be in complete darkness for one hour
  Arms: Light exposure darkness

SUMMARY:
Monochromatic light creates longitudinal chromatic aberration, with short wavelength blue light forming a focal point in front of the retina and long wavelength red light forming a focal point behind the retina. The investigators hypothesize that such chromatic aberrations, induced by exposure to red or blue LED lights, will cause the choroid behind the retina to respond to bring the image into focus by modulating its thickness, either thickening in the case of blue light or thinning in the case of red light. The magnitude and direction of this response is difficult to predict as previous studies have shown opposite findings in non-human primates and rodents. Furthermore, the investigators hypothesize that exposure to red or blue light will induce changes in how the pupil responds to light, because the cells in the eye that are involved in pupil control are most sensitive to blue light.

DETAILED DESCRIPTION:
Ambient light exposure is associated with choroid thickness and eye growth. The spectral composition of light, which has been shown to play a role in eye growth, can differentially regulate changes in choroid thickness by forming a focal point either in front of the retina in the case of short wavelength blue light or behind the retina in the case of long wavelength red light. In addition, melatonin suppression and the pupil light response, specifically, that driven by the intrinsically photosensitive retinal ganglion cells (ipRGCs), are most sensitive to short wavelength blue light. Therefore, the role of the wavelength of light on eye growth may involve ipRGC activity. As such, it is relevant to determine whether exposure to monochromatic light will alter choroidal thickness, ipRGC activity and melatonin levels.

The purpose of this study is to compare the short-term changes in choroid thickness, melatonin concentration, and the ipRGC-driven pupillary light response following one hour of light therapy with either short wavelength blue light or long wavelength red light. It has previously been shown that a one week period of daily morning light therapy produces a short term increase in choroid thickness throughout the day. Therefore, the investigators hypothesize that one hour of morning light therapy with short wavelength blue light will result in different effects in the changes in choroid thickness, melatonin levels, and the ipRGC-driven pupillary light response compared to one hour of morning light therapy with long wavelength red light.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-64
* must be able to comply with the experimental protocol, including collecting saliva and being present for the experiment in the lab on four separate occasions.
* must be willing to abstain from the use of sleep aids 12 hours prior to and for the duration of the study.
* must also be willing to abstain from alcohol and caffeinated beverages (coffee, espresso, energy drinks) or foods enriched with caffeine, such as power bars, the morning of and during each of the four experimental sessions.

Exclusion Criteria:

* age < 18 or >64 years old
* not willing to collect a saliva sample or be present in the lab on four separate occasions.
* ocular disease that may affect retinal light levels and function (e.g. glaucoma, significant cataract, etc.)
* use of prescription or over-the-counter medications known to affect sleep and cortisol levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Choroidal Thickness | one hour
  The choroid will be imaged with OCT to determine choroidal thickness
Pupil response | one hour
  The pupil response will be measured before and after one hour to see if exposure to light affects the diameter

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston College of Optometry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lou L, Ostrin LA. Effects of Narrowband Light on Choroidal Thickness and the Pupil. Invest Ophthalmol Vis Sci. 2020 Aug 3;61(10):40. doi: 10.1167/iovs.61.10.40. PMID 32832970
- See also: published manuscript — https://pubmed.ncbi.nlm.nih.gov/32832970/